CLINICAL TRIAL: NCT07174050
Title: Comparison of the King Vision Channeled Videolaryngoscope and Conventional Laryngoscopy for Endotracheal Intubation Time in Novice Users: A Prospective, Randomised Controlled Trial
Brief Title: King Vision vs Macintosh Laryngoscopy for Intubation Time in Novice Users
Acronym: KVVL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hitit University (Other)
Collaborators: Izmir City Hospital (Other Government)
Responsible Party: Principal Investigator, Murat KAYKAC, M.D., Izmir City Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KINGVISON1; 2018/5 (Other: Health Sciences University Izmir Bozyaka Training and Research Hospital Clinical Research Ethical Committee)
Record Dates: First submitted 2025-09-08; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Airway Management; Endotracheal Intubation; Tracheal Intubation, Elective Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group K (Experimental): Channelled blade of KVVL
  Interventions: Device: King Vision Channeled Video Laryngoscope
- Group M (Active Comparator): Macintosh laryngoscope
  Interventions: Device: Macintosh Laryngoscopy

INTERVENTIONS:
Device: King Vision Channeled Video Laryngoscope — King Vision Videolaryngoscope (KVVL) is one of the new indirect laryngoscopes with disposable (either with channeled or non-channeled) blades .Both designs include an anti-fog lens coating . The channelled KVVL has a rigid blade with an integrated channel for introducing the endotracheal tube. The height and width of the standard non-channeled and channeled blades are 13 mm and 26 mm vs 18 mm and 29 mm, respectively. The KVVL has a unique design and high-quality image . It has a camera that enables a clear view of the glottis. It is a solid, portable, battery-operated device with an organic LED display for video laryngoscopy . It allows better glottis visualization and Cormack Lehane score than DL. Compared with Airtraq, the KVVL has wide field of view (160° vs 80° respectively) and potentially shortens the time to tracheal intubation .
  Arms: Group K
Device: Macintosh Laryngoscopy — In clinical practice, direct laryngoscopy (DL) with either a curved (Macintosh) or straight (Miller) blade is a well-known and reliable technique in the hands of an experienced operator.
  Arms: Group M

SUMMARY:
This study evaluated two different devices used for placing a breathing tube (endotracheal intubation) in adult patients undergoing elective surgery. The aim was to compare the King Vision videolaryngoscope, which has a camera and a guiding channel for the tube, with the traditional Macintosh laryngoscope, which allows doctors to look directly at the vocal cords. The study focused on how long it takes to successfully insert the tube, the need for additional maneuvers during the procedure, and the overall success rate of first attempts. The procedures were performed by novice operators under supervision.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years old) scheduled for elective surgery under general anesthesia requiring orotracheal intubation
* American Society of Anesthesiologists (ASA) physical status I-II
* Mallampati airway classification I-II
* Written informed consent obtained from the patient

Exclusion Criteria:

* Predicted or known difficult airway: Mallampati III-IV, inter-incisor distance <2.5 cm, thyromental distance <6 cm, limited cervical spine mobility
* History of difficult intubation or need for awake/rapid-sequence intubation
* Upper airway pathology (tumour, trauma, infection), limited mouth opening, or craniofacial anomalies
* Emergency surgery, high aspiration risk, or full stomach
* Severe cardiopulmonary instability (e.g., shock, severe hypoxaemia)
* Pregnancy or breastfeeding
* BMI >35 kg/m² (if your protocol excludes obesity; remove if not applicable)
* Participation refusal or inability to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Time to successful endotracheal intubation (seconds) | During intubation (intraoperative period, approximately 1-2 minutes)
  Measured from insertion of the laryngoscope blade between the patient's incisors until removal of the blade after correct placement of the endotracheal tube, confirmed by capnography.

CONTACTS AND LOCATIONS:
Locations (1):
- Izmir City Hospital, Izmir, Turkey (Türkiye)